CLINICAL TRIAL: NCT01031745
Title: Contingency Management in the Delivery of HAART to Drug Users in Chennai, India
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: YR Gaitonde Centre for AIDS Research and Education (Other)
Responsible Party: Principal Investigator, Gregory M. Lucas, Professor of Medicine, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01-DA018577-S3; R01DA018577 (NIH)
Record Dates: First submitted 2009-12-12; First posted 2009-12-15 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: HIV; Substance Abuse, Intravenous
Keywords: Complementary Therapies; Drug Users
MeSH Terms: conditions — Substance Abuse, Intravenous; Drug Misuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contingency (Experimental)
  Interventions: Behavioral: Contingency
- Control (Active Comparator)
  Interventions: Other: Prize bowl drawings

INTERVENTIONS:
Behavioral: Contingency — Participants are provided a non-monetary incentive for achieving particular tasks between study visits. Tasks include initiation of HAART, timely refill of medications from the government ART centers, suppression of HIV RNA
  Arms: Contingency
Other: Prize bowl drawings — Control participants receive counseling and referral, but no incentives for engagement in HIV care. At study visits they are eligible to receive "bonuses" through prizebowl drawings to offset the inability to earn incentives.
  Arms: Control

SUMMARY:
Drug use (DU) is a major risk factor for HIV infection in many regions of the world. However, as highly active antiretroviral therapy (HAART) has been rolled out in South and South East Asia, less than 2% of individuals initiated on HAART were drug users (DUs) or former DUs, despite the fact that approximately 20% of HIV infections in the region are ascribed to DU. India is home to about 2.4 million HIV-infected individuals. Though, injection drug users contribute to only about 3% of all HIV infections in India; it is estimated that there are between 168,000 and 1.1 million DUs in India with HIV prevalence about 30%. Novel approaches are needed to engage disenfranchised populations in HIV care in lower and middle income countries, where the burden of HIV disease is growing. Incentive-based strategies (or contingency management) have been shown to be effective in reducing illicit drug use, smoking cessation, and weight loss. Short-term pilot studies have also shown that incentive-based strategies can improve electronically-monitored rates of adherence to HAART in the US, and a recent study in Africa showed that a small incentive approximately doubled the rate that individuals returned to learn the results of their HIV test. However, to date there is no experience with the use of incentive-based interventions to improve engagement into care and risk-reduction among out-of-care HIV-infected DUs in developing world settings. The investigators propose to conduct pilot randomized trial comparing a voucher incentive strategy to a control condition to improve engagement in HIV care and HIV treatment outcomes among out-of-care, treatment-eligible, HIV-infected DUs in Chennai, India. Subjects in the incentive arm will be eligible to earn incentive vouchers for 1) initiating HAART at a government-sanctioned HIV treatment clinic, 2) adherence to scheduled follow-up visits at the HIV clinic, and 3) achieving suppression of HIV RNA. Subjects will be enrolled from a mature research venue in Chennai, YR Gaitonde Centre for Substance Abuse-related Research (YRGCSAR), which focuses the epidemiology and natural history of HIV in DUs. Preliminary data from this pilot study will be used to inform the design of a phase-III study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Provide written informed consent
* Provide a history of injection or non-injection drug use in prior 30 days
* Documented evidence of HIV infection
* Be ART naïve (by self-report)
* Satisfy Indian National Guidelines for initiation of HAART (any of the following)

  * Absolute CD4+ count < 200 cells/ µl
  * AIDS-defining illness with any CD4+ count
  * Absolute CD4+ count between 200 - 350 cell/ µl with HIV-related symptoms

Exclusion Criteria:

* Indicates an intention to migrate in the next 12 months
* Any medical or psychiatric condition that the study physician believes to be a contraindication to study participation.
* Enrolled in another HIV treatment program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Time to initiation of HAART | 12 months

SECONDARY OUTCOMES:
Attendance at HIV treatment visits | 12-months
HAART possession ratio (a surrogate of medication adherence based on pharmacy fill data) | 12-months
Proportion with HIV RNA < 400 copies/mL at 6- and 12-months | 12-month
Changes in absolute CD4 count from baseline at 6- and 12-months | 12-months

CONTACTS AND LOCATIONS:
Locations (1):
- YR Gaitonde Centre for Substance Abuse-Related Research (YRGCSAR), Chennai, Tamil Nadu, India

REFERENCES:
- [Result] Solomon SS, Srikrishnan AK, Vasudevan CK, Anand S, Kumar MS, Balakrishnan P, Mehta SH, Solomon S, Lucas GM. Voucher incentives improve linkage to and retention in care among HIV-infected drug users in Chennai, India. Clin Infect Dis. 2014 Aug 15;59(4):589-95. doi: 10.1093/cid/ciu324. Epub 2014 May 6. PMID 24803381